CLINICAL TRIAL: NCT04391491
Title: Neuregulin-1 in Patient With Different Forms of Cardiovascular Diseases: a Pilot Study
Acronym: NRG-1-CVDs
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: Universiteit Antwerpen (Other); University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 03-19 13022019
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Microvascular Angina; Pulmonary Hypertension; Heart Failure With Reduced Ejection Fraction
Keywords: Neuregulin-1; Microvascular Angina,Heart Failure,Pulmonary Hypertension
MeSH Terms: conditions — Microvascular Angina; Hypertension, Pulmonary; Fibromatosis, Gingival, 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples for analysis of neuregulin-1β, NT-proBNP, biomarkers of inflammation and fibrosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Heart failure with preserved ejection fraction: Patients of both sexes and > 18 years with a confirmed diagnosis of HFpEF (Symptoms of HF (NYHA II-IV); LVEF >50%; Elevated levels of natriuretic peptides (NT-pro BNP > 300 pg/ml in sinus rhythm, >600 pg/ml in AF);Relevant structural heart disease (Left ventricle hypertrophy (LVH) and/or Left atrium enlargement (LAE); left atrial volume index (LAVI) >34 mL/m2 or a left ventricular mass index (LVMI) =115 g/m2 for males and =95 g/m2 for females)
  Interventions: Diagnostic Test: Neuregulin-1β level in plasma
- Microvascular angina: Patients of both sexes and > 18 years with a confirmed diagnosis of MVA (Angina-like chest pain: signs of exercise-induced ischemia (ST-depression on exercise ECG (>1 mm down-sloping or rectilinear ST-segment depression in >2 leads)); No fixed stenosis (>50%) in epicardial coronary arteries or branches at baseline coronary arteriography)
  Interventions: Diagnostic Test: Neuregulin-1β level in plasma
- Pulmonary hypertension: Patients of both sexes and > 18 years with a confirmed diagnosis of secondary PH due to left heart disease (Left ventricular systolic dysfunction, left ventricular diastolic dysfunction, Valvular disease, Congenital/acquired left heart inflow/outflow obstruction and congenital cardiomyopathies) or chronic thromboembolic pulmonary hypertension defined by echo when peak tricuspid regurgitation velocity =2.8 m/s and presence of other echo 'PH signs'
  Interventions: Diagnostic Test: Neuregulin-1β level in plasma
- Heart failure with redused ejection fraction: Patients of both sexes and > 18 years with a confirmed diagnosis of HFrEF (Symptomatic HF (NYHA class II-IV), left ventricular ejection fraction ≤ 35% (at any time in the past))
  Interventions: Diagnostic Test: Neuregulin-1β level in plasma

INTERVENTIONS:
Diagnostic Test: Neuregulin-1β level in plasma — Peripheral blood will be collected after randomization (plus or minus 3 days), the plasma will be assayed for neuregulin-1b, biomarkers of inflammation and fibrosis, NTproBNP

SUMMARY:
This is an observational study of Neuregulin-1 (NRG-1) plasma levels in patients with different forms of cardiovascular disease including microvascular angina (MVA), heart failure with preserved ejection fraction (HFpEF), as well as, heart failure with reduced ejection fraction (HFrEF) and pulmonary hypertension (PH). Investigators intend to identify cardiovascular diseases which are characterized by increased circulating NRG-1, considered to be a biomarker of therapeutic potential of NRG-1. Participants will undergo blood sampling over 3 days following randomisation. Patients demographics and clinical characteristics will be recorded and their associations with NRG-1 will be analysed.

DETAILED DESCRIPTION:
NRG-1 is a paracrine growth factor with physiological actions in the cardiovascular system which is primarily expressed by the endothelium of coronary microvessels. NRG-1 is a natural paracrine agonist of the ErbB4 receptor. The NRG-1/ErbB4 system is activated in chronic heart failure (HF) and some other chronic diseases, exerting disease mitigation and regenerative effects. Recombinant NRG-1 (rhNRG-1) is developed as a drug for HFrEF. Both the preclinical and clinical data (phase II and III clinical trials) have demonstrated the favourable effects of NRG-1 treatment on the heart. rhNRG-1 effectively enhances the heart function and reverses the remodelling of the left ventricle. The levels of circulating NRG-1 were found to correlate with outcomes in Stage III and IV CHF. NRG1 appeared to be potentially protective Therefore, NRG-1 concentrations are considered to be a biomarker of the therapeutic potential of NRG-1. However, little is known about the role of the NRG-1 pathway in other cardiovascular diseases (CVDs). This observational study is intended to identify CVDs which are characterized by an increase in NRG-1 levels for better positioning the NRG-1 treatment in heterogeneous field of CVDs. Based on preclinical data, investigators assume that plasma NRG-1 will be altered in patients with microvascular angina, pulmonary hypertension, and HFpEF and HFrEF.

The study intends to enroll twenty patients for each of the 4 study groups and 20 healthy controls. We will compare the NRG-1 protein levels in patients and of age-matched healthy subjects. Participants will undergo a blood sampling after randomization (+ 3 days) and a 12 month follow up to assess the outcomes. Demographics, clinical characteristics, laboratory values including biomarkers of inflammation and fibrosis, NTproBNP, along with transthoracic echo findings and outcomes will be recorded. After the active phase of the research is done, we are planning to proceed to observation of the prospective group of patients to verify the endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Confirmed diagnosis of HFpEF (Symptoms of HF (NYHA II-IV); LVEF >50%; Elevated levels of natriuretic peptides (NT-pro BNP > 300 pg/ml in sinus rhythm, >600 pg/ml in AF);Relevant structural heart disease (Left ventricle hypertrophy (LVH) and/or Left atrium enlargement (LAE); left atrial volume index (LAVI) >34 mL/m2 or a left ventricular mass index (LVMI) =115 g/m2 for males and =95 g/m2 for females)
* Confirmed diagnosis of MVA (Angina-like chest pain: signs of exercise-induced ischemia (ST-depression on exercise ECG (>1 mm down-sloping or rectilinear ST-segment depression in >2 leads)); No fixed stenosis (>50%) in epicardial coronary arteries or branches at baseline coronary arteriography)
* Confirmed diagnosis of PH (PH due to left heart disease (Left ventricular systolic dysfunction, Left ventricular diastolic dysfunction, Valvular disease, Congenital/acquired left heart inflow/outflow obstruction and congenital cardiomyopathies); Chronic thromboembolic pulmonary hypertension; Peak tricuspid regurgitation velocity =2.8 m/s and presence of other echo 'PH signs')
* Confirmed diagnosis of HFrEF (Symptomatic HF (NYHA class II-IV), left ventricular ejection fraction ≤ 35% (at any time in the past))

Exclusion Criteria:

* Patients with hypertrophic cardiomyopathy, rheumatic heart disease, constrictive pericarditis, significant valvular pathological change or congenital heart diseases
* Primary pulmonary artery hypertension
* Acute MI in the last 3 months
* Unstable angina
* Chronic heart failure patients with acute decompensation in the last 1 month (symptoms and signs suggest worsening chronic heart failure and may require intravenous drug therapy)
* Cardiac surgery or cerebrovascular accident within the recent six months
* Severe hepatic or renal dysfunction
* Severe nervous system diseases
* History of any malignancy or suffering from cancer
* Lack of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of pulmonary hypertension, microvascular angina, heart failure with preserved ejection fraction or heart failure with reduced ejection fraction as defined by the diagnostic criteria in respective ESC guidelines
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
NRG-1 plasma concentrations | up to 3 days
  Peripheral blood will be collected after randomization (plus or minus 3 days) in vacuum tubes containing EDTA. Blood samples will be centrifugated within 30 minutes of collection. Then plasma will be separated and procced for NRG-1 measurement using the R&D ELISA (R&D cat# DY377)

SECONDARY OUTCOMES:
Correlations between NRG-1 and NTproBNP, biomarkers of inflammation and fibrosis | 14 days
  Correlations between NRG-1 and NTproBNP, biomarkers of inflammation and fibrosis will be assessed with suitable correlation analyses depending on normality of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Shchendrygina, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Anastasia Shchendrygina, Moscow, Russia

REFERENCES:
- [Background] De Keulenaer GW, Feyen E, Dugaucquier L, Shakeri H, Shchendrygina A, Belenkov YN, Brink M, Vermeulen Z, Segers VFM. Mechanisms of the Multitasking Endothelial Protein NRG-1 as a Compensatory Factor During Chronic Heart Failure. Circ Heart Fail. 2019 Oct;12(10):e006288. doi: 10.1161/CIRCHEARTFAILURE.119.006288. Epub 2019 Oct 14. PMID 31607147